CLINICAL TRIAL: NCT07187882
Title: Autologous Non-cultured Epidermal Cell Suspension Transplantation in the Treatment of Vitiligo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Ding Xiaolan, Associate Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDL2023-04
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Vitiligo
Keywords: non cultured epidermal cell suspension; vitiligo; autologous
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NCES (Experimental)
  Interventions: Procedure: Autologous Non-cultured Epidermal Cell Suspension transplantation

INTERVENTIONS:
Procedure: Autologous Non-cultured Epidermal Cell Suspension transplantation — 1. Thin split thickness skin grafts were taken from the donor site (anterolateral thigh) after application of topical anaesthesia under complete aseptic precautions.
  2. The cell suspension was prepared by the cell sorting kit (Primcell, Jiangsu Repatec Life Science Co.,Ltd).
  3. Then the recipient skin was uniformly dermabraded using an electrical dermabrader set at 10,000 to 20,000 rpm until punctate bleeding points appeared.
  4. The cell suspension was applied onto the dermabraded recipient area.
  5. The recipient site was then fixed firmly with dressings and elastic bandage. The dressings were removed 10 days after transplantation.

SUMMARY:
To observe the long-term efficacy and safety of autologous non cultured epidermal cell suspension transplantation in the treatment of vitiligo, analyze the correlation between cell density, type, and postoperative efficacy and prognosis, and providing a basis for clinical application.

DETAILED DESCRIPTION:
1. Patient recruitment Inclusion criteria：

1. Patients diagnosed as vitiligo, according to the "Vitiligo Diagnosis and Treatment Consensus (2021 edition)
2. Segmental and unclassified vitiligo stable for 6 months, Non-segmental vitiligo stable for 1 year and resistant to medication and phototherapy
3. BSA≥5%
4. Sign the informed consent and be willing to undergo surgical treatment
5. 8-65 years old, both genders Exclusion criteria：

1) Severe visceral or infectious disease not suitable for surgical treatment 2) Tendency toward keloid formation 3) Coagulation defects 4) Unable to complete follow-up on time 2. Non-cultured epidermal cell suspension transplantation procedure

1. Thin split thickness skin grafts of about one-tenth of the recipient area were taken from the donor site(anterolateral thigh)after aseptic precautions.
2. The suspension for non-cultured epidermal cell suspension transplantation was prepared by the cell sorting kit (Primcell, Jiangsu Repatec Life Science Co.,Ltd).
3. The recipient site was cleaned with 75% alcohol and anesthetized by applying topical compound lidocaine cream for 45 to 60 minutes. Then the recipient skin was uniformly dermabraded using an electrical dermabrader set at 10,000 to 20,000 rpm until punctate bleeding points appeared. Dermabrasion was performed 0.5 mm beyond the margin of the recipient area to minimize the perigraft halo of depigmentation.
4. The cell suspension was applied onto the dermabraded recipient area. The recipient site was then fixed firmly with 4 layers of dressing. From the inner to the outer layer, these dressings were: non adherent wound dressing , paraffin-embedded gauze, dry gauze, and elastic bandage. The dressings were removed 10 days after transplantation.

3. Postoperative Follow-Up All patients returned to the hospital for follow-up examinations at 2 weeks, 1month, 2 months, 3 months, 4 months, 5 months and 6 months after transplantation.

The repigmentation was graded based on the percentage of the area of repigmentation as poor (less than 25%), good (26%-50%), very good (51%-75%), or excellent (more than 75%).

The melanin index (MI) and erythema index (EI) of the recipient sites were measured using a Mexameter MX18 (Courage 1Khazaka Electronic GmbH, Koln, Germany). The relative MI (RMI) and relative EI (REI) were calculated as the ratio of the MI or EI of the recipient sites relative to the symmetrical control skin region.

4. Laboratory Tests The cell number and vitality of the suspension was determined by an automatic intelligent cell counter. The flow cytometry was used to analyze the cell types.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as vitiligo, according to the "Vitiligo Diagnosis and Treatment Consensus (2021 edition)
* Segmental and unclassified vitiligo stable for 6 months, Non-segmental vitiligo stable for 1 year and resistant to medication and phototherapy
* BSA≥5%
* Sign the informed consent and be willing to undergo surgical treatment
* 8-65 years old, both genders

Exclusion Criteria:

* Severe visceral or infectious disease not suitable for surgical treatment
* Tendency toward keloid formation
* Coagulation defects
* Unable to complete follow-up on time

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Repigmentation rate | 2 weeks, 1month, 2 months, 3 months, 4 months, 5 months and 6 months after transplantation
  The repigmentation rate depends on the percentage of repigmentation area /recipient area*100%. The extent of repigmentation was devided as poor (less than 25%), good (26%-50%), very good (51%-75%), or excellent (more than75%).

SECONDARY OUTCOMES:
Relative Melanin Index | 2 weeks, 1month, 2 months, 3 months, 4 months, 5 months and 6 months after transplantation
  The melanin index (MI) of the recipient sites were measured using a Mexameter MX18 (Courage 1Khazaka Electronic GmbH, Koln, Germany). The relative MI (RMI) and were calculated as the ratio of the MI of the recipient sites relative to the symmetrical control skin region
Relative erythema index | 2 weeks, 1month, 2 months, 3 months, 4 months, 5 months and 6 months after transplantation
  The erythema index (EI) of the recipient sites were measured using a Mexameter MX18 (Courage 1Khazaka Electronic GmbH, Koln, Germany). The relative EI (REI) were calculated as the ratio of the EI of the recipient sites relative to the symmetrical control skin region

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No